CLINICAL TRIAL: NCT05762965
Title: Effect of Galacto-oligosaccharides (GOS) on Faecal Gut Microbiota in Adult Women
Acronym: Denali
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 6239229900
Record Dates: First submitted 2023-02-08; First posted 2023-03-10 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Microbial Colonization
Keywords: galacto-oligosaccharides; prebiotics; microbiota
MeSH Terms: conditions — Communicable Diseases | interventions — 4'-galactooligosaccharide

STUDY DESIGN:
Intervention Model Description: The study applies a randomized, parallel, double-blind design of 6 weeks
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GOS 1 (Experimental): Galacto-oligosaccharide
  Interventions: Dietary Supplement: GOS 1
- GOS 2 (Experimental): Galacto-oligosaccharide
  Interventions: Dietary Supplement: GOS 2

INTERVENTIONS:
Dietary Supplement: GOS 1 — 1 sachet each morning
  Other Names: galacto oligosaccharide
  Arms: GOS 1
Dietary Supplement: GOS 2 — 1 sachet each morning
  Other Names: galacto oligosaccharide
  Arms: GOS 2

SUMMARY:
Within the Denali study the effect of 3 weeks intervention with GOS on the abundance of Bifidobacterium in faecal samples will be investigated.

DETAILED DESCRIPTION:
This randomized, parallel, double-blinded intervention study of 6 weeks will include 88 females, who will consume GOS for three consecutive weeks. Faecal samples will be collected at several time points to measure microbiota composition.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy women
* Aged between 40 - 70 year
* Body Mass Index (BMI) between 18.5 - 30 kg/m2

Exclusion Criteria:

* Having a gastro-intestinal disease, such as celiac disease, Crohn's disease, Ulcerative colitis, or diagnosed irritable bowel syndrome;
* Having a history of intestinal surgery that might interfere with study outcomes. This does not include an appendectomy or cholecystectomy;
* Diagnosed with diabetes mellitus;
* Use of medication that may influence the study results, such as laxatives, lactase preparations, metformin, antibiotics, proton pomp inhibitors, antipsychotics, NSAID's (judged by our research physician);
* Self-perceived and diagnosed constipation;
* Having a food allergy to cow's milk or being lactose intolerant;
* Self-reported slimming, medically prescribed or other diets
* Reported weight loss or weight gain of >5kg in the month prior to screening
* Use of (foods with) pre-, pro-, syn- and/or postbiotics* (should be stopped at least 4 weeks before the start of the study), or other supplements that can influence the study results (to be determined by the medical investigator);
* History of side effects with the use of prebiotic supplements
* Use of antibiotic treatment less than 3 months before start of the study
* Pregnant or lactating (or having the wish to become pregnant during the study period, self-reported);
* Not able to comply with study procedures;
* Use of drugs (should be stopped at least 4 weeks before the study);
* Alcohol intake ≥7 glasses of alcoholic beverages per week, on average
* Participation in another clinical trial at the same time;
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research or employee of FrieslandCampina R&D.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Enrollment: 88 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
faecal abundance of Bifidobacterium | At week -3 (start control)
  faecal abundance of Bifidobacterium.
faecal abundance of Bifidobacterium | At week 0 (end control)
  faecal abundance of Bifidobacterium.
faecal abundance of Bifidobacterium | At week 3 (end intervention)
  faecal abundance of Bifidobacterium.

SECONDARY OUTCOMES:
Faecal microbiota composition | At week -3 (start control)
  Gene-based microbiota profiling of faecal samples
Faecal microbiota composition | At week 0 (end control)
  Gene-based microbiota profiling of faecal samples
Faecal microbiota composition | At week 3 (end intervention)
  Gene-based microbiota profiling of faecal samples

CONTACTS AND LOCATIONS:
Overall Officials: Maartje van den Belt, Msc, Principal Investigator — Wageningen Food and Biobased Research
Locations (1):
- Wageningen University & Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Looijesteijn E, Schoemaker MH, van den Belt M, Hester ER, Kortman GAM, Viskaal-van Dongen M, Nauta A. A double-blind intervention trial in healthy women demonstrates the beneficial impact on Bifidobacterium with low dosages of prebiotic galacto-oligosaccharides. Front Nutr. 2024 Aug 19;11:1440319. doi: 10.3389/fnut.2024.1440319. eCollection 2024. PMID 39224188